CLINICAL TRIAL: NCT02403258
Title: The Effect and Safety of Plum-blossom Needle for Tourette Syndrome: a Randomized Controlled Trial
Brief Title: The Effect and Safety of Plum-blossom Needle for Tourette Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yu Jinna, Attending doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014S298
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Tourette Syndrome
Keywords: acupuncture; plum-blossom needle; tourette syndrome; randomized controlled trial
MeSH Terms: conditions — Tourette Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plum-blossom needle group (Experimental): Patients randomized into this group will receive plum-blossom needle as treatment. DU 20, DU 16, GB 20, EX-HN5, BL 15, BL 18, BL 23 will be selected as acupoints. Each point will be tapped gently one by one by plum blossom needle until the skin get slightly redness. The treatments will be given two sessions per week, consistently for 12weeks (24 sessions in all).
  Interventions: Other: Plum-blossom needle group
- HRT group (Active Comparator): Patients randomized into this group will receive habit reversal training (HRT) as treatment. Habit reversal training will consist of the following 4 parts: (1) self-monitoring, (2) competing responses, (3) relaxation training and (4) contingency management. The training will be given weekly in the 12 weeks (totally 12 sessions) by a special rehabilitation therapist, first two sessions 1.5 h, and remaining sessions 1 h for each treatment.
  Interventions: Behavioral: HRT group

INTERVENTIONS:
Other: Plum-blossom needle group — Plum-blossom needle is a method of shallow insertion with multiple needles. It is made of five or seven stainless steel needles arranged in a pattern like the shape of plum blossom, thus named as 'plum-blossom needle'. Plum-blossom needle treat diseases by tapping specific skin areas or acupoints according to different illness based on the theory of meridian.
  Other Names: acupuncture; plum-blossom needle
  Arms: Plum-blossom needle group
Behavioral: HRT group — HRT consisted of (1) self-monitoring, (2) competing responses, (3) relaxation training, (4) contingency management.
  Arms: HRT group

SUMMARY:
To evaluate the effect and safety of plum-blossom needle for Tourette syndrome.

DETAILED DESCRIPTION:
This is a randomized, controlled trial with two parallel arms. A total of 60 patients will be randomly allocated into the plum-blossom needle group (n=30) and the habit reversal training (HRT) group (n=30). 12-week treatment will be given to all patients of each group, follow-up will be made at the 12th week after treatment. The primary outcome measure will be the mean change from baseline in the total tic score on the Yale Global Tic Severity Scale (YGTSS) at the 12th week. Secondary outcome measures will include the mean changes in score of YGTSS, TS Clinical Global Impression Scale (CGI) and the Children and Adolescents' Quality of Life Scale from baseline at other time. Safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association (DSM-IV) for TS.
2. Aged 7 to 18.
3. Agree to participate in the trial and sign written informed consent by both guardians and subjects.

Exclusion Criteria:

1. Having severe problem in heart, liver or kidney, or having hyperthyroidism.
2. After evaluated by psychiatrists based on the Kiddie-Sads-Present and Lifetime Version, those who are associated with co-morbid conditions such as mental retardation, pervasive developmental disorder, schizophrenia, mania episode, bipolar disorder, anxiety and depression and specific learning disorder will be excluded.
3. Tics symptoms caused by some drugs.
4. Currently receiving any other form of pharmacological or non-pharmacological treatment for their Tourette syndrome.
5. Patients with a history of psychotropic substance or alcohol use during the 3 months preceding screening.
6. Patients with a history of nonresponsiveness to HRT or participating in another clinical trial.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change of YGTSS score from baseline at the 12th week | baseline, week 12
  the symptom scale used in this trial will be the Yale Global Tic Severity Scale. (YGTSS).

SECONDARY OUTCOMES:
change of YGTSS score from baseline at other point times | baseline, week 4, week 8, week 24.
  this outcome will be measured by the Yale Global Tic Severity Scale.
CGI score | week 4, week 8, week 12, week 24.
  this outcome will be measured by the TS Clinical Global Impression Scale (CGI).
change of quality of life from baseline | baseline, week 12, week 24.
  this outcome will be measured by the Children and Adolescents' Quality of Life Scale (CAQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Jinna Yu, Ph.D, Study Chair — Guang'an Men Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We haven't get consent from patients to share their individual data with other researchers.

REFERENCES:
- [Derived] Yu J, Ye Y, Li S, Liu J, Zhai Y, Zhang M, Liu Z. The effectiveness and safety of plum-blossom needle therapy for Tourette syndrome: study protocol for a randomized controlled trial. Trials. 2015 Jul 29;16:320. doi: 10.1186/s13063-015-0873-0. PMID 26220439